CLINICAL TRIAL: NCT04032639
Title: Chronic Stress, Cognition, and Food Cue Reactivity in Prader-Willi Syndrome: A Magnetoencephalography Study
Brief Title: Stress and Brain Response Using MEG in PWS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Holland Bloorview Kids Rehabilitation Hospital (Other); University of Western Ontario, Canada (Other)
Responsible Party: Principal Investigator, Jill Hamilton, Principal Investigator, The Hospital for Sick Children
Other Study IDs: 1000061983
Record Dates: First submitted 2019-07-11; First posted 2019-07-25 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Prader-Willi Syndrome
Keywords: Prader-Willi Syndrome; Magnetoencephalography; Food Cue Reactivity; Stress
MeSH Terms: conditions — Prader-Willi Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — A fasting blood sample will be collected to measure glucose, insulin, cortisol, active peptide YY, and active ghrelin
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prader-Willi Syndrome: 24 children and adolescents (7-16 years) with diagnosed Prader-Willi Syndrome will be recruited
- Controls: 24 children and adolescents (7-16 years) without diagnosed Prader-Willi Syndrome will be matched for age, sex, and BMI-percentile to the Prader-Willi group

SUMMARY:
Individuals with Prader-Willi Syndrome (PWS) have increased hunger and food seeking behaviour, as well as learning (cognitive) challenges. In addition, some patients with PW been shown to have low cortisol production, particularly in stressful situations. However, research examining how hormonal, cognitive, and psychological factors are interrelated PWS is limited. To address this gap in knowledge, the goal of this project is to understand how changes in brain regions involved in controlling food intake and cognitive processes are related to changes in hormones regulating appetite, the stress hormone cortisol, and performance on neuropsychological tests.

DETAILED DESCRIPTION:
Prader-Willi Syndrome (PWS) is characterized by hyperphagia, although the degree of food seeking can vary between individuals. This behaviour may be moderated by hormonal, neurocognitive, and psychological factors; however, data assessing these factors in an integrated fashion is scarce. The proposed research will address and identify relationships between three major challenges in PWS: 1) dysregulated feeding behaviour, 2) cognitive performance, and 3) chronic stress. The investigators will measure brain response to food cues, during a cognitive task, and at rest using magnetoencephalography (MEG) in adolescents with PWS and BMI-matched controls. This is an innovative design as previous studies in this population used only functional magnetic resonance imaging (fMRI) to examine food cue reactivity, which does not directly measure neuronal activity and lacks temporal-sensitivity. In contrast, MEG directly records neural firing and combines high spatial resolution with exquisite temporal resolution, allowing us to measure functional connectivity between brain regions. Importantly, MEG is also patient-friendly with fewer contraindications than MRI. To assess cognitive function, the investigators will utilize gold-standard neuropsychological measures, as well as emotional and social behavioural functioning. Lastly, the investigators will assess hair cortisol, which is a reflection of long term, month-by-month cortical exposure. This new area of research will explore neurobiological and cognitive mechanisms controlling feeding behaviour in PWS.

ELIGIBILITY:
Inclusion Criteria:

* Genetically diagnosed PWS (study population)
* Adolescents matched for age, sex, and BMI-percentile (controls)

Exclusion Criteria:

* Past or current history of alcoholism or consistent drug use
* Current untreated major psychiatric illness as defined by the DSM-V criteria
* Medications that decrease alertness (that cannot be held on the days of testing)
* History of recent major head trauma
* Current pregnancy
* Diagnosis of diabetes
* Current or recent smoker (i.e. >2 cigarettes/week during past year)
* History of metal in body (shrapnel, metal slivers, unremovable metal adornments, clips, top braces, pacemaker)
* Use of glucocorticoid medications

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Prader-Willi Syndrome (PWS) is characterized by hyperphagia, although the degree of food seeking can vary between individuals. The characteristic endocrine and metabolic dysfunction in PWS is indicative of abnormalities in the hypothalamus, and other brain systems. In addition to the hyperphagia and risk for obesity, anxiety is a prominent feature of PWS
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2019-05-30 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Neuronal activity during the food cue reactivity task | 2 years
  To compare neuronal activity between PWS and controls during the food cue task

SECONDARY OUTCOMES:
Relationships between appetite hormone response and neuronal activity during the food cue task | 2 years
  To compare how appetite hormones correlate with neuronal activity in PWS compared to controls
Relationships between cortisol and neuronal activity during the food cue reactivity task | 2 years
  To compare how stress correlates with neuronal activity in PWS compared to controls
Neuronal activity during the emotional processing task | 2 years
  To compare neuronal activity between PWS and controls during the emotional processing task
Neuronal activity during resting state | 2 years
  To compare neuronal activity between PWS and controls during resting state
Neuronal activity during the response inhibition task | 2 years
  To compare neuronal activity between PWS and controls during the response inhibition task
Relationships between neuropsychological function and neuronal activity during the emotional processing task | 2 years
  To compare how neuropsychological function correlate with neuronal activity in PWS compared to controls
Relationships between cortisol and neuronal activity during the emotional processing task | 2 years
  To compare how stress correlates with neuronal activity in PWS compared to controls

OTHER OUTCOMES:
Relationships between neuropsychological function and neuronal activity during the food cue reactivity task | 2 years
  To compare how neuropsychological function correlate with neuronal activity in PWS compared to controls
Relationships between neuropsychological function and neuronal activity during the response inhibition task | 2 years
  To compare how neuropsychological function correlate with neuronal activity in PWS compared to controls

CONTACTS AND LOCATIONS:
Overall Officials: Jill Hamilton, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada